CLINICAL TRIAL: NCT05608434
Title: Development of Virtual Reality-based Interventions to Strengthen Cognitive Skillsets Related to Attention Deficit Hyperactivity Disorder (ADHD): A Pilot Phase I and Randomized Controlled Phase II Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000744; 000744-M
Record Dates: First submitted 2022-11-04; First posted 2022-11-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11-19

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Smart Games; Neurodevelopmental; Virtual Reality; fMRI; Cognitive Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Floreo VR group (Experimental): This group will undergo up to 20 daily sessions (20 minutes each) of the Floreo VR training.
  Interventions: Behavioral: Floreo Virtual Reality application

INTERVENTIONS:
Behavioral: Floreo Virtual Reality application — Floreo VR is a novel VR-based cognitive training therapy for ADHD. It incorporates multiple learning modules, each of which targets a neuropsychological domain relevant to ADHD (inhibitory control, working memory, temporal processing, processing speed). The demands of the training intervention adapt to the subject s practice-driven improvements in performance. Specifically, when the subject is deemed to perform adequately well at a given level of difficulty, the training adapts by presenting a more challenging difficulty. This adaptation to the subject s performance is designed to allow for continued incremental improvements in the trained domains. The VR games take place in a spaceship themed environment. The VR training is designed to be used at home, under the supervision of a parent.

SUMMARY:
Background:

Children with attention deficit hyperactivity disorder (ADHD) often have cognitive problems. It may be hard for them to control their behaviors, concentrate for long periods, or make decisions. This can affect their education, friendships, and daily life. Virtual reality-based games may help improve cognitive skills in children with ADHD. It may also help change how the brain functions.

Objective:

To see if virtual reality-based games help improve thinking skills and brain function in children with ADHD.

Eligibility:

Children aged 8 to 16 years with ADHD.

Design:

We will first do a pilot study, meaning that everyone will receive the games. If this is successful, we will then conduct a randomized controlled trial, meaning that some participants will be randomly assigned to the full version of the games and some will be randomly assigned to a limited version. Participants will be screened. Their physical and mental health, medical and family history, and intellectual and emotional development will be evaluated. They will have tests of their mood, memory, attention, thinking, and behavior. Blood or saliva may be collected. Participants may have an MRI scan of the brain.

Participants will receive a set of virtual reality games. The set includes 4 different games all played using a virtual reality headset. The participant will play the games for 20 minutes 5 days a week for 4 weeks.

The parent or caregiver will start each game using an iPad. Each of the games is designed to help the participant practice specific cognitive skills. These include inhibition control, processing speed, temporal information processing, and working memory.

Participants will have interviews each week. They will answer questions about motion sickness, eye strain, headache, and any other side effects, as well as number of game sessions played.

Blood or saliva tests and the MRI may be repeated after the last game session. For the pilot, participants will have a final interview at the study end. For the full trial, a 1-month follow-up visit will be done by telehealth.

DETAILED DESCRIPTION:
Study Description: This study will be a randomized double-blind placebo-controlled trial examining the efficacy of a novel virtual reality (VR) adaptive cognitive training intervention for youth with ADHD in improving symptoms of inattention relative to a non-adaptive training control intervention. Prior to the main randomized trial, a proof-of concept open-label pilot study will assess the safety, tolerability, usability, feasibility, credibility and treatment expectancy of the intervention. It will also provide an initial assessment of the efficacy on the intervention in improving inattention symptoms and neuropsychological performance.When these parameters are met, the pilot will be complete and the RCT will begin.

Objectives:

Primary Objective: Examine the efficacy of the Floreo VR intervention in improving symptoms of inattention in children/adolescents with ADHD.

Secondary Objectives: Examine the efficacy of the VR intervention in improving neuropsychological performance in four cognitive domains pertinent to ADHD.

Pilot Study Objective: Assess the safety, tolerability, usability, feasibility, credibility and treatment expectancy of the VR intervention. Provide an initial open-label assessment of the efficacy of the intervention.

Endpoints:

Primary Endpoint: The primary endpoint of the main trial is to investigate whether the intervention decreases symptoms of inattention as assessed using the ADHD Rating Scale-5 for Children and Adolescents (ADHD-RS-5).

A secondary aim of the main study is to investigate whether the intervention brings about improvements in performance on four neuropsychological performance indices. These are stop signal reaction time on the Stop Signal task (inhibitory control), visuospatial working memory as determined using number of correct responses on the Dot Matrix task, a composite measure of temporal deviation on a Temporal Reproduction task, and the number of correct responses on the NIH Toolbox Pattern Comparison Processing Speed Test.

Pilot intervention Endpoints: Responses to structured interview items on safety, tolerability, usability, credibility and treatment expectancy of the intervention. Reports of adverse events will be used to assess safety. Feasibility will be assessed using participation and compliance rates. Usability will also be assessed using a System Usability Scale. Open-label assessments of efficacy will also be performed, using the ADHD-RS-5 inattention subscale. Secondary endpoints for the pilot study are the same as for the main study.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate, an individual must meet all of the following criteria:

1. Children must provide informed assent and parents must provide informed consent to participate in the study.
2. Any sex assigned at birth, or race/ethnicity.
3. Aged between 8 and 16 years of age, including all months leading up to age 17.
4. Meets diagnosis for ADHD, predominately inattentive or combined presentations, or a specified presentation of having prominent symptoms of inattention that are impairing in two or more settings (but not numerous enough to meet a diagnosis of inattentive or combined presentation).
5. Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study.
6. For the Pilot only: If treated for ADHD with psychostimulants, willing to withdraw medication three days prior to baseline assessments and to stay off medication until completion of the post-intervention assessment. Not receiving any other psychotropic medication for at least 30 days prior to baseline assessment.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Cognitively not capable of performing study procedures. Indications of a lack of cognitive capacity could include a known IQ under 70, or a history from the screening interview that implies global intellectual disabilities (e.g., placement in a school for children with intellectual disability etc.)
2. History of severe migraines, vertigo, epilepsy (with the exception of febrile seizures), or serious balance disorders.
3. Impairments in uncorrected visual acuity that would interfere with engagement with the VR training.
4. Known to be pregnant.
5. Psychotic disorders (including schizophrenia, psychosis not otherwise specified), current substance dependence. Other psychiatric disorders elicited on the interview are not considered exclusionary provided that ADHD is considered to be one of the dominant sources of impairment for the child.
6. Considered a suicide risk as determined during the clinical interview at baseline.
7. Any other medical or psychiatric condition that in the opinion of the PI may confound study data/assessments (e.g., limitations in mobility that would render the VR headset unusable).
8. Recent (within three months) treatment with other cognitive training interventions (e.g., Cogmed) for ADHD.
9. The VR equipment produces excessive discomfort to the child in the opinion of the PI (e.g., including participants with small interpupillary distances (IPD) that are only able to see blurry images on the VR headset, or children showing signs of undue neck and upper body strain or fatigue while trying the headset).
10. For the main trial only: Certain psychotropic medications classes that are likely to interfere with the completion of the intervention are exclusionary: antipsychotics, mood stabilizers (lithium, valproate, lamotrigine, gabapentin). Medications for ADHD will not be considered as exclusionary. This includes psychostimulants, atomoxetine, alpha 2 adrenergic agonists. Antidepressant and anxiolytic medication will also not be exclusionary if they are deemed not to not interfere with study procedures
11. For the main trial only: Prior use of Floreo s products including but not limited to their ADHD cognitive training application.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
ADHD-RS-5 inattention sub-scale. | within one month of the end of VR training
  The ADHD-RS-569 is a rating scale based on the diagnostic criteria for ADHD as described in the DSM-5. Inattention symptoms are one of two key symptom domains for ADHD, and the target of the present intervention.

SECONDARY OUTCOMES:
Number of correct responses on the NIH Toolbox Pattern Comparison Processing Speed Test. | within one month of the end of VR training
  Computerized neuropsychological assessment of processing speed
Number of correct responses on the Dot Matrix task | within one month of the end of VR training
  Computerized neuropsychological assessment of working memory
Temporal deviation on a temporal reproduction task | within one month of the end of VR training
  Computerized neuropsychological assessment of motor-timing
Stop signal reaction time on the Stop Signal task (inhibitory control) | within one month of the end of VR training
  Computerized neuropsychological assessment of inhibitory control

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified medical information will be placed in a NIH repository (e.g., Biomedical Translational Research Information System (BTRIS)) in accordance to NIH policies. We will also share genomic and phenotypic data in controlled access databases such as dbGAP (database of Genotypes and Phenotypes). Other databases may be used as approved by NIH for the sharing of de-identified data.
Supporting Information: Study Protocol
Time Frame: The timeline for data sharing will follow the NHGRI Genomic Data Sharing Policy. Currently data is deposited following IRB review once the study data collection is complete and the data has undergone quality control steps.
Access Criteria: Access requests for specific research purposes using NIH controlled-access data are reviewed by NIH Data Access Committees (DACs).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000744-M.html